CLINICAL TRIAL: NCT04821167
Title: Safety and Efficiency of Laparoscopic Management of Intra-canalicular (Emergent) Testis
Acronym: LapUDT
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: dr. Muhammad Abdelhafez Mahmoud, MD (Other)
Responsible Party: Sponsor-Investigator, dr. Muhammad Abdelhafez Mahmoud, MD, Lecturer of pediatric surgery, Al-Azhar Faculty of Medicine, Al-Azhar University
Organization: Al-Azhar University (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: Al-AzharLapUDT
Record Dates: First submitted 2021-03-24; First posted 2021-03-29 (Actual); Last update posted 2021-03-29 (Actual); Status verified 2021-03

CONDITIONS: Testes Undescend
Keywords: Laparoscopic,; orchiopexy,; intracanalicuar testes,; peeping testes
MeSH Terms: conditions — Cryptorchidism | interventions — Orchiopexy

STUDY DESIGN:
Intervention Model Description: This is a prospective study conducted to evaluate the safety and efficiency of laparoscopic orchiopexy of intra-canalicular (emergent/peeping) testis.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Laparoscopic orchiopexy for intra-canalicular (emergent or peeping) testis (Other): This is a prospective study conducted on male children with intermittent palpable (peeping) UDT to evaluate the safety and efficiency of laparoscopic orchiopexy of intra-canalicular (emergent or peeping) testis.
  Interventions: Procedure: laparoscopic orchiopexy for intra-canalicular testis

INTERVENTIONS:
Procedure: laparoscopic orchiopexy for intra-canalicular testis — laparoscopic orchiolysis of abnormal fibrous attachments and then lap assisted transcrotal fixation of the testis in subdartos pouch for intra-canalicular testis

SUMMARY:
Undescended testes (UDTs) are a relatively common finding in pediatrics with prevalence about 1-2% in newborns. Upon discovering a non-intrascrotal testis, it is important to determine whether the testis is palpable or non-palpable (1). A canalicular or 'emergent' testis may be impalpable initially and may be appear when it is 'milked' out of the inguinal canal (where it is concealed from detection) indicating that 15 to 40% of cryptorchidism are viable peeping/canalicular testis.

The laparoscopic approach for treating canalicular undescended testes offers many advantages over open inguinal orchiopexy. The laparoscopic technique maintains the integrity of the inguinal canal anatomy and eliminating the need to divide the epigastric vessels during dissection. The ability to dissect the testicular vessels at a higher extent would increase the vessel length available to lower the testis without strain.

* This is a prospective study will be conducted at Department of Pediatric Surgery, MCH hospital, Bisha, Saudia Arabia and Pediatric surgery Department , Al-Azhar University hospitals, Cairo, Egypt, from January 2019 to October 2020 to evaluate the safety and efficiency of laparoscopic orchiopexy of intracanalicular testis.
* Patients' age and laterality will be reported. Evaluation will be done for the operative difficulties, intraoperative complications, operative time and early postoperative complications.

Testicular site, size and vascularity will be evaluated by ultrasonography at 6th month post operatively. Also, cosmetic results will be evaluated by obtaining the parent's questioners at post-operative OPD clinic visits.

- Laparoscopic orchiopexy for management of inguinal canalicular undescended testes is a safe, effective, and less invasive, without disturbance of inguinal canal anatomy, with better cosmetic results.

DETAILED DESCRIPTION:
Aim of the study:

Herein, the study aims to evaluate the laparoscopic procedure for management of canalicular testis regarding operative safety, efficacy and post-operative outcomes.

Brief review of literature:

* Different management modalities for intra-canalicular (emergent) testes in male children (open surgery, Laparoscopy).
* Advantages of laparoscopic orchiopexy for intra-canalicular (emergent) testes.

Patients and Methods:

This is a prospective study, will be conducted out at pediatric surgery tertiary centers (Maternity & Children's Hospital in Bisha, KSA and Al-Azhar University hospitals in Cairo, Egypt) on pediatric patients presenting at the pediatric surgery OPD clinic by intra-canalicular (emergent/peeping) testes in the period from January 2019 to October 2020. Enrolled patients will be managed by laparoscopic orchiopexy. All patients enrolled in the study will give a written informed consent. The study will be approved by the Institutional Review Board and ethics committee of the hospitals. The main objective is to assess safety and efficacy of laparoscopic orchiopexy for intra-canalicular (emergent/peeping) testes in male patients.

Institutes of the study:

A multicenter study at Pediatric Surgery Departments, Maternity & Children's hospital in Bisha, KSA and Al-Azhar University hospitals in Cairo.

Number of cases: Sixty two male children. Time frame: period of 1.10 years.

Ethical Consideration:

The protocol will be discussed and approved for clinical study by the Ethical Research Committee at MCH at Bisha, KSA, and other participating hospitals. The procedures and the aim of the study will be clearly explained to the patient and the family. A written informed consent will be obtained before enrollment of the patients into the study. The family refusal to give consent for laparoscopic management is respected but does not deprive the patient from getting open orchiopexy.

Preoperative preparation:

Proper examination done for patients using flat and frog leg position with gentile squeezing of testis down, proved by preoperative inguinoscrotal ultrasonography.

Follow-up:

Patients will be reviewed at the OPD clinic. Patients who could not attend the clinic will be contacted by phone. Postoperative Doppler ultrasonography will be done to assess testicular size and vascularity. Questionnaire will be obtained from the parents to assess their cosmetic satisfaction.

Statistical analysis:

It will be performed with IBM SPSS Statistics for Windows, Version 23.0. Armonk, NY: IBM Corp. Data will be presented as mean, standard deviation, number & percentage, using Chi-squared test (X2) for qualitative data. The significance level will be set at P > 0.05.

- Discussion will focus on laparoscopic management of intra-canalicular (emergent) testes. The results obtained from this study will be compared with each other and with that reported in the literature. The discussion will focus on operative details, operative time, results, & complications.

It will compare results of this study with the results of others. Discussion will determine the most accurate management modality for intra-canalicular (emergent) testes in male children which offers the best outcome and least morbidity.

ELIGIBILITY:
Inclusion Criteria:

* All children diagnosed as intra-canalicular (emergent/ peeping) testes

Exclusion Criteria:

* Patients above 14 years of age,
* with retractile testes,
* with retractile testes that were distal to the external ring and
* with nonpalpable testes

Ages: 8 Months to 48 Months | Sex: Male | Healthy Volunteers: No
Age Groups: Child
Gender Based: Yes — Male children with intra-canalicular (emergent/ peeping) testes
Enrollment: 62 (Actual)
Dates: Start 2019-01-01 (Actual); Primary Completion 2020-04-20 (Actual); Study Completion 2020-10-31 (Actual)

PRIMARY OUTCOMES:
Patients' age (in months) | 2 years
  Patients' age
Patients' weight (in kilograms) | 2 years
  Patients' weight
Side of affected testis (number of cases) | 2 years
  The side of the affected testis

SECONDARY OUTCOMES:
Operative time (in minutes) | 1 day (day of surgery)
  Operative time
Testicular size (in cubic milliliters) | 2 years
  Testicular size measurement by ultrasonography
Testicular site (in centimeters) | 2 years
  Testicular distance from the mid-scrotum point to evaluate that it remained in the scrotum or re-ascended
Parents' satisfaction (percent of each satisfaction grade) | 2 years
  Parents' satisfaction questionnaire
Period of follow-up (in months) | 2 years
  Follow-up period

CONTACTS AND LOCATIONS:
Locations (1):
- Mohammad Alsayed Daboos, Cairo, Egypt

IPD SHARING:
Plan to Share IPD: Yes
Data are available for other researchers including methodology, figures, tables, results, and philosophy of discussion and the value this study add to the literature
Supporting Information: Study Protocol, SAP, ICF
Time Frame: October 2020 till indefinitely
Access Criteria: after the article became accepted and available online.